CLINICAL TRIAL: NCT05805111
Title: CERAB - Prospective, Non-Randomised Clinical Trial to Investigate the BeGraft Aortic Stent Graft System and the BeGraft Peripheral Stent Graft System Treating Aortic-iliac Occlusive Disease With CERAB
Brief Title: Prospective, Non-Randomised Clinical Trial to Investigate the BeGraft Aortic Stent Graft System and the BeGraft Peripheral Stent Graft System Treating Aortic-iliac Occlusive Disease
Status: Recruiting | Type: Observational
Sponsor: Marc Bosiers, MD (Other)
Responsible Party: Sponsor-Investigator, Marc Bosiers, MD, Dr., FCRE (Foundation for Cardiovascular Research and Education)
Organization: FCRE (Foundation for Cardiovascular Research and Education) (Other)
Other Study IDs: FCRE-200622
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Aorto-iliac Occlusive Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: endovascular intervention — Covered Endovascular Reconstruction of Aortic Bifurcation (CERAB) is a new, minimally invasive technique, for treating extensive and/or recurrent aorto-iliac occlusive disease. The technique rebuilds the diseased aortic bifurcation and iliac arteries through the use of stent-grafts introduced through the groin or arm arteries.

SUMMARY:
This is a prospective, multi-center, investigational study to evaluate safety and performance of the BeGraft Aortic balloon expandable covered Stent Graft System and the BeGraft Peripheral balloon expandable covered stent Graft System (Bentley InnoMed GmbH, Hechingen, Germany) implanted as covered stents in CERAB procedures (Covered Endovascular Reconstruction of Aortic Bifurcation) for extensive aorto-iliac occlusive disease.

The objective of this clinical investigation is to evaluate the safety and performance of the BeGraft Aortic covered stent Graft System & the BeGraft Peripheral covered stent Graft System (Bentley Innomed, Hechingen, Germany) in CERAB configuration (Covered Endovascular Reconstruction of Aortic Bifurcation) for Aorto-iliac Occlusive Disease.

ELIGIBILITY:
General Inclusion criteria

1. Patient has been identified with an chronic aorto-iliac occlusive lesion, with clinical necessity for treatment.
2. The patient has been diagnosed with symptomatic peripheral artery disease, defined by Rutherford Becker Classification score 2 to 5.
3. Patient has a projected life-expectancy of at least 24 months.
4. Patient is ≥18 years old.
5. Patient is willing/capable and provides written consent to participate to the trial and confirmed to attend the expected follow-up visits.

Angiographic inclusion criteria:

1. Patient's anatomy is eligible for CERAB treatment, without the need for chimneys and can be treated with a Ø 12 mm BGA.
2. The aorto-iliac lesion begins at least 1 cm below the patent renal arteries without a need for treatment.
3. A maximum of 3 BeGraft Peripheral (Ø 7 or 8 mm) per limb in the iliac artery can be used. In case a Ø 7 mm is used to extend, the overlapping end must be post-dilated to ensure proper flow.
4. The target lesion has angiographic evidence of stenosis >50% or occlusion.
5. Patient's common femoral artery and deep femoral artery are patent.

General Exclusion criteria:

1. Patient is currently participating in another interventional drug trial or device trial that has not completed the entire follow up period.
2. Patient has planned any surgical intervention/procedure, that is not related to the study procedure, within 30 days after the study procedure.
3. Patient had a Myocardial infarction or stroke within a period of 3 months prior to the study procedure.
4. Patient had surgery (e.g. bypass surgery or stenting) in target vessels previously.
5. Patient has an acute severe systemic infection at time of screening or in period of 30 days prior to screening.
6. Patient has fresh thrombus at time of screening or in period of 14 days prior to screening.
7. Patient has a CERAB procedure that is staged.
8. Female patient with childbearing potential not taking adequate contraceptives.
9. Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated.
10. Patients with known hypersensitivity to the stent material (L605) and/or PTFE.
11. Patients who are placed in an institution due to an institutional or court order.
12. An aneurysm in the abdominal aortic and iliac segments where CERAB will be placed is present.
13. Patient has or had aortic coarctation.
14. Patient had aortic injury/trauma related interventions previously.
15. Patient had suprarenal/visceral segment reconstructions previously.

Angiographic exclusion criteria

1. Failure of recanalization
2. A relevant accessory renal artery (>3 mm) in the infrarenal aorta is present, that might be occluded during the procedure.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aorto-iliac occlusive disease, who have been diagnosed by means of Rutherford Becker Classification between 2 and 5.
Sampling Method: Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Freedom from clinically-driven target lesion revascularization | at 12 months after procedure
  Freedom from clinically-driven target lesion revascularization (CD-TLR) at 12 months, defined as freedom from repeat endovascular revascularization to maintain or re-establish patency within the treated lesion.
Incidence of Serious Adverse Device Effects | at 12 months after procedure
  Incidence of Serious Adverse Device Effects (SADE) and procedure related Serious Adverse Events (SAE) at 12 months follow up.

SECONDARY OUTCOMES:
Technical success rate after procedure | at procedure
  Technical success rate after procedure defined as successful introduction and deployment of the study devices BeGraft Aortic covered stent Graft System & the BeGraft Peripheral covered stent Graft System (Bentley Innomed, Hechingen, Germany) for CERAB procedures
Freedom for conversion to open surgical repair | at 30 days post-procedure, 6-, 12-, and 24-months
  Freedom for conversion to open surgical repair of the target lesion.
Patency rate of the target vessel | at 30 days post-procedure, 6-, 12-, and 24-months
  Patency rate of the target vessel (primary, primary assisted and secondary).
Time to re-vascularization/re-intervention | at 30 days post-procedure, 6-, 12-, and 24-months
  Time to re-vascularization/re-intervention
Patient reported outcomes | at 30 days post-procedure, 6-, 12-, and 24-months
  Patient reported outcomes at 30 days post-procedure, 6-, 12-, and 24-months compared to pre-procedure
Clinical success at every follow up visit | at 30 days post-procedure, 6-, 12-, and 24-months
  Clinical success at every follow up visit, defined as an improvement of Rutherford classification of one class or more compared to the pre-procedure Rutherford classification
Hemodynamic improvement | at 30 days post-procedure, 6-, 12-, and 24-months
  Hemodynamic improvement defined as increase in Ankle Brachial Index (ABI) of at least 0.10 compared to baseline ABI (pre-procedure) at 30 days post-procedure, 6-, 12-, and 24-months.
Safety endpoints | at 30 days post-procedure, 6-, 12-, and 24-months
  1. Incidence of Serious Adverse Device Effects (SADE) and procedure related Serious Adverse Events (SAE)
  2. 30-day mortality.
  3. Overall survival rate
  4. Incidence of Major Adverse Events

CONTACTS AND LOCATIONS:
Locations (15):
- Germany (9):
  - Sankt Gertrauden-Krankenhaus, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - University Medical Center Goettingen, Göttingen
  - Universitätsklinikum Heidelberg, Heidelberg
  - Marienhospital Lünen, Lünen
  - St. Franziskus-Hospital GmbH, Münster
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
  - Uniklinikum Regensburg, Regensburg
  - Klinikum der Landeshauptstadt Stuttgart gKAöR, Stuttgart
- Netherlands (6):
  - Noordwest Ziekenhuisgroep Alkmaar, Alkmaar
  - Ziekenhuis Rijnstate Arnhem, Arnhem
  - Martini Ziekenhuis, Groningen
  - UMCG Groningen, Groningen
  - Maastricht UMC+, Maastricht
  - HMC (Haaglanden Medisch Centrum), The Hague

IPD SHARING:
Plan to Share IPD: No